CLINICAL TRIAL: NCT05656430
Title: Internet-based Cognitive Behavioral Therapy for Psychological Symptoms Related to the COVID-19 Pandemic Remaining After Societal Opening
Brief Title: ICBT for Psychological Symptoms Related to the COVID-19 Pandemic Remaining After Societal Opening
Acronym: PCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PostCoronaCope
Record Dates: First submitted 2022-12-16; First posted 2022-12-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depression Symptoms; Anxiety Symptoms
Keywords: COVID-19; Corona; Postpandemic; Internet-based cognitive behavioral therapy (ICBT); Internet intervention; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: After recruitment finished, participants will be randomized to either intervention condition (treatment group) or control condition (wait list). Participants in the control group will receive the same treatment once the intervention group has finished the treatment and outcome measures has been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Eight weeks of individually tailored ICBT, were participants receives in total 8 modules out of 20 possible depending on their current problems and described situation with weekly support by a therapist.
  Interventions: Behavioral: Internet-based Cognitive Behavioral Therapy
- Control group (No Intervention): The control group is a wait-list control condition. Participants are instructed to wait. After the treatment group has finished their treatment and post-treatment measures has been collected, the control group receive the same treatment as the treatment group got.

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavioral Therapy — Intervention based on cognitive behavioural therapy principles and adapted to the coronavirus pandemic situation. The 20 modules that the intervention consists of include psycho-educational texts as well as examples and exercises.
  Arms: Treatment group

SUMMARY:
This study aim to investigate the effects of internet-based cognitive behavioral therapy (ICBT) addressing psychological symptoms related to the COVID-19 pandemic and its consequences that remain after societal opening. The target group is adults (18 years or older) who still experience psychological symptoms related to the pandemic and the ICBT consists of eight modules during eight week with weekly support by a therapist. ICBT will be compared to a wait-list control condition. Participants will be recruited in Sweden with nationwide recruitment.

DETAILED DESCRIPTION:
The study is a randomized controlled trial about the effects of ICBT regarding psychological symptoms related to the COVID-19 pandemic and its consequences remaining after societal opening. Primary outcome measures are depression symptoms (measured with Beck Depression Inventory-II) and anxiety symptoms (measured with Generalized Anxiety Disorder-7). Other outcome measures used will for example be about stress symptoms, sleep problems, post traumatic stress symptoms and quality of life.

Because of uncertainties about the psychological effects of COVID-19 pandemic, a transproblematic individually tailored treatment will be used that has been tested in several previous trials and adapted for addressing problems related to the pandemic and its consequences. The study (nor the recruitment within it) has not a focus on whether people have or have not been infected by the COVID-19 virus.

ELIGIBILITY:
Inclusion Criteria:

* Experience mental health problems related to the COVID-19 pandemic and/or its consecuences, which are still experienced as a problem (when the pandemic is not considered as dangerous to the society)
* 18 years or older
* Adequate ability to speak, read and write in Swedish
* Having access to the internet and a smartphone, computer or other device

Exclusion Criteria:

* Severe psychiatric or somatic issues that makes participation harder or impossible (which can include the diagnosis postcovid)
* Ongoing addiction
* Acute suicidality
* Other ongoing psychological treatment
* Recent (within the past 3 months) changes in the dose of psychotropic medication or planned change during the treatment weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Becks Depression Inventory-II | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of depressive symptoms. Range for the total sum is between 0 and 63 with a higher score indicating a higher level of depressive symptoms. Clinical ranges for minimal, mild, moderate and severe major depressive disorder are considered to be 0-13, 13-19, 20-28, and 29-63 points respectively.
Generalized Anxiety Disorder-7 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of anxiety symptoms and worry. When summing the points of the seven first questions, the scores are interpreted as mild, moderate and severe anxiety symptoms at 5-10, 11-15 and above 15 respectively.

SECONDARY OUTCOMES:
Percieved Stress Scale-14 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A questionnaire that aims to measure symptoms of stress. I contains 14 items that are scored on a range betewwn 0 (never) to 4 (very often). The total score range is between 0-56 and a higher score reflects higher levels of perceived stress.
Insonnia Severity Index | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of insomnia severity and symptoms of disordered sleep. Norm score ranges include low likelihood of sleep problems (0 to 7 points), some sleep problems (8 to 14 points), moderate sleep problems (15 to 21 points), severe sleep problems (22 to 28 points).
Short Health Anxiety Inventory-14 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of health anxiety, short version, with 14 items which are answered on a scale 0-3. This gives a total scare range of 0-42, where 0-14 indicate low probability of health anxiety, 15-17 is a grey zone and points over 18 indicates high probability for health anxiety.
Alcohol Use Disorder Identification Test | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. 10 items and scores ranging from 0-40 with higher scores indicating a higher level of alcohol use.
Karolinska Exhaustion Disorder Scale 9 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A questionnaire aiming to measure fatigue and exhaustion. Maximum score is 54 and people scoring higher than 18 points are considered as being at risk for exhaustion syndrome.
Impact of Event Scale-6 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A short version of Impact of Event Scale-R (IES-R), which assesses subjective distress caused by potentially traumatic events. It yields a total score between 0-24 with a higher score indicating more severe distress caused by the traumatic events.
UCLA loneliness scale 3 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A short version of the UCLA loneliness scale, aiming to measure with three questions, for example "How often do you feel left out?" and are answered on a scale ranging from 1 (hardly ever) to 3 (often). People who gets the score 3-5 have been grouped as not lonely, while score 6-9 has been grouped as lonely.
Brunnsviken Brief Quality of Life Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of quality of life with a total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.
The Cognitive Failures Questionnaire | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  The measure contains 25 questions and are aiming to measure the experience of the frequency of misstakes one does in the every day life because of problems with attention, memory, and emotion regulation. Maximum score are 100, where higher score mirrors experienced problems to a greater extent.
InCharge Financial Distress/Financial Well-Being Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A measure aiming to measure distress related to the individual's economic situation. It contains of eight questions where the respondent gets to answer on a scale from 1 to 10.

OTHER OUTCOMES:
Knowledge test | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Knowledge test about cognitive behavior therapy and how strategies in cognitive behavior therapy can be applied in every day situations. It consists of 16 questions and the respondent gets three answer options while one of the alternatives are correct. The respondent also gets to answer how confident he/she is about the answer (I'm guessing, I'm pretty certain, I'm quite certain).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden